CLINICAL TRIAL: NCT00002682
Title: CURRENT PRACTICE STUDY OF ANTIBIOTIC TREATMENT OF GASTRIC MALT LYMPHOMA
Brief Title: Antibiotic Therapy and Antacids in Patients With Malt Lymphoma of the Stomach
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPPDM95-084; P30CA016672 (NIH); MDA-CPPDM-95084; NCI-T95-0003D; CDR0000064361 (Other: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-06-10 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Lymphoma
Keywords: Antibiotic Treatment; Gastric Malt Lymphoma; stage I marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell, Marginal Zone | interventions — Amoxicillin; bismuth subsalicylate; Clarithromycin; Metronidazole; Omeprazole; Tetracycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antibiotic Treatment (Experimental)
  Interventions: Drug: Amoxicillin; Drug: Bismuth Subsalicylate; Drug: Clarithromycin; Drug: Metronidazole Hydrochloride; Drug: Omeprazole; Drug: Tetracycline Hydrochloride

INTERVENTIONS:
Drug: Amoxicillin
Drug: Bismuth Subsalicylate
Drug: Clarithromycin
Drug: Metronidazole Hydrochloride
Drug: Omeprazole
Drug: Tetracycline Hydrochloride

SUMMARY:
RATIONALE: Antibiotic therapy and antacids are used to treat Helicobacter pylori infection of the stomach. These treatments may also have an effect on gastric MALT lymphoma of the stomach.

PURPOSE: Phase II trial to study the effectiveness of antibiotic therapy with amoxicillin, clarithromycin, tetracycline, and metronidazole plus antacids in patients with MALT lymphoma of the stomach.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the response of gastric lymphoma of mucosa-associated lymphoid tissue (MALT) to treatment for Helicobacter pylori infection with antibiotics (amoxicillin, clarithromycin, tetracycline, and metronidazole) and with gastric acid inhibitors (omeprazole and bismuth subsalicylate). II. Correlate response with endoscopic tumor grade and clinical and pathological parameters. III. Assess the incidence of H. pylori infection in patients with gastric MALT lymphoma.

OUTLINE: All patients are treated on Regimen A; those receiving tetracycline on Regimen A are switched to Regimen B for their second course; those receiving amoxicillin for their first course receive tetracycline for their second course. Regimen A: Antibiotic Therapy with Gastric Acid Inhibition. Amoxicillin (or Tetracycline in penicillin-allergic patients); Clarithromycin; with Bismuth Subsalicylate; Omeprazole. Regimen B: Antibiotic Therapy with Gastric Acid Inhibition. Tetracycline; Metronidazole, METRO, NSC-50364; with Bismuth Subsalicylate; Omeprazole.

PROJECTED ACCRUAL: 75 patients will be entered over 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Suspected gastric lymphoma or documented gastric lymphoma of mucosa-associated lymphoid tissue (MALT) that is stage IE Gastric MALT lymphoma with perigastric lymph nodes identified on endoscopic ultrasound eligible at MDACC and Houston VA Medical Center only No indication for expeditious treatment with chemotherapy, radiotherapy, or surgery based on clinical condition, underlying illness, or tumor stage

PATIENT CHARACTERISTICS: Age: 18 to 80 Performance status: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No contraindication to endoscopy or biopsy No pregnant or nursing women Adequate contraception required of fertile patients

PRIOR CONCURRENT THERAPY: No concurrent chemotherapy or radiotherapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 1995-08-10 (Actual); Primary Completion 2001-10-08 (Actual); Study Completion 2001-10-08 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Response to Antibiotic Treatment of Gastric Malt Lymphoma | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Steinbach, MD, PhD, Study Chair — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - University of Texas - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org